CLINICAL TRIAL: NCT00990457
Title: Two Diets With Exercise in Abdominal Obesity: Cardiovascular Effects
Brief Title: Evaluating the Effects Two Diets Combined With Exercise in Persons With Abdominal Obesity (The SHAPE5 Study)
Acronym: SHAPE5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kerry Stewart, Professor of Medicine, National Heart, Lung, and Blood Institute (NHLBI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 682; 5R01HL092280 (NIH); 1R01 092280
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Overweight; Obese; Sedentary; Abdominal Obesity
Keywords: Exercise; Weight loss diet; Obesity; Overweight; Abdominal obesity; Cardiovascular function; Body composition
MeSH Terms: conditions — Overweight; Obesity; Sedentary Behavior; Obesity, Abdominal; Motor Activity | interventions — Diet, Reducing; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-carbohydrate Diet Plus Exercise (Active Comparator): Participants will follow a low-carbohydrate weight loss diet plus participate in a supervised exercise training program for 6 months.
  Interventions: Behavioral: Weight Loss Diets Plus Exercise
- Low-Fat, Low-Calorie Diet Plus Exercise (Active Comparator): Participants will follow a low-calorie, low-fat weight loss diet plus participate in a supervised exercise training program for 6 months.
  Interventions: Behavioral: Weight Loss Diets Plus Exercise

INTERVENTIONS:
Behavioral: Weight Loss Diets Plus Exercise — The weight loss diet will be either a low-carbohydrate diet or a low-fat, low-calorie diet. All participants will also be enrolled in a supervised exercise program.
  The supervised exercise training sessions will take place three times a week for 6 months. Each session will last 1 to 1 ½ hours and will include aerobic exercise and weight training.

SUMMARY:
Abdominal obesity, which is affected by a lack of physical activity and excess weight, put people at an increased risk of cardiovascular disease. This study will compare the effects of two different dietary approaches to weight loss, each combined with exercise, for their effects on cardiovascular factors that are early predictors of future cardiovascular disease in overweight and obese people with excessive weight around their waist. The two diets are a low-carbohydrate versus a more traditional low-fat, low calorie diet.

DETAILED DESCRIPTION:
Abdominal obesity is a condition that is largely influenced by a poor diet and physical inactivity. This condition has adverse effects on heart and blood vessel structure and function, including left ventricular diastolic dysfunction, endothelial vasodilator dysfunction, and increased vascular stiffness, each of which increase the risk of cardiovascular disease. Reducing the amount of calories consumed and increasing physical activity are both important factors for losing weight, increasing fitness, and improving blood glucose control. However, little research has been conducted on comparing different diet approaches combined with exercise for their effects on general and abdominal obesity, fitness, heart and blood vessel structure and function, and heart disease risk factors. The purpose of this study is to determine whether people who follow low-carbohydrate diet or a low-fat, low-calorie diet, each combined with a supervised experience similar improvements in cardiovascular and in body composition and health.

This study will enroll people who are overweight or obese and abdominal obesity, defined as a waist to hip ratio greater than 1, or a waist size of 40" or greater in men or 35" or greater in women. Participants will attend baseline study visits and complete blood pressure measurements; muscle strength measurements; a treadmill test to evaluate cardiovascular fitness; an echocardiogram to obtain images of the heart; tests to measure blood vessel function; a dual energy x-ray absorptiometry (DEXA) scan to measure body fat, muscle tissue, and bone density; questionnaires to assess physical activity levels, quality of life, and mood; and a blood collection. A portion of blood will be stored for future genetic testing. Women will also provide a urine sample for pregnancy testing. Participants will also keep a food diary for 3 days. Participants will then be randomly assigned to either a low-carbohydrate or a low-fat, low-calorie weight loss diet, each combined with a supervised exercise program. . The exercise program will be done three times a week for 6 months. Each session will last 1 to 1 ½ hours and will include aerobic exercise and weight training.

All participants will attend study visits with a dietitian for weight loss counseling and monitoring once a week during Months 1 and 2, and every other week in Months 3 through 6. At each of these visits, participants' weight will be measured.

At the end of Month 6, all participants will attend a study visit for repeat baseline testing. In addition, there will another test for vascular function, BP, weight, and waist and hip measurements at the time a participant loses ten pounds.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30-65 years old
* Body mass index (BMI) of 25-42 kg/m^2
* Waist of 35 inches or greater in women and 40 inches or greater in men; or, a
* Waist-hip ratio greater than 1.

Exclusion Criteria:

* Currently smokes
* History or evidence of cardiovascular disease or other major chronic illness
* Currently exercising regularly or following a weight loss diet
* Diabetes
* Uncontrolled high blood pressure
* Any illness that would prevent participation in a moderate-intense exercise program
* Pregnant
* Substance abuse

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Cardiovascular structure and function | Measured at 6 months

SECONDARY OUTCOMES:
Body composition | Measured at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry J Stewart, EdD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States